CLINICAL TRIAL: NCT01688999
Title: A Phase II Study of Cabozantinib (XL184) in Patients With Advanced/Metastatic Urothelial Carcinoma
Brief Title: Cabozantinib for Advanced Urothelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Andrea Apolo, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120205; 12-C-0205
Record Dates: First submitted 2012-09-14; First posted 2012-09-20 (Estimated); Results first posted 2020-10-06 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-09

CONDITIONS: Urothelial Carcinoma; Urethral Neoplasms; Urinary Bladder Neoplasms; Kidney Neoplasms
Keywords: Kidney Cancer; Tyrosine Kinase Inhibitor; Bladder Cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urethral Neoplasms; Urinary Bladder Neoplasms; Kidney Neoplasms | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cabozantinib (Experimental): Administered orally at a dose of 60 mg once daily on each day of a 28-day cycle.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — 60 mg by mouth (PO) daily each 28 day cycle. Treatment continues until toxicity or disease progression.
  Other Names: Cometriq

SUMMARY:
Background:

- Cabozantinib is a drug that slows the growth of blood vessels that feed tumors. It is approved for medullary thyroid cancer. However, studies have shown that prostate and ovarian tumors respond to it. Researchers want see if cabozantinib can be a safe and effective treatment for urothelial cancer.

Objectives:

- To test the safety and effectiveness of cabozantinib for advanced urothelial cancer.

Eligibility:

- Individuals at least 18 years of age who have advanced urothelial cancer that has not responded to standard treatments.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. Tumor tissue samples will also be collected. Imaging studies will also be performed.
* Participants will take cabozantinib by mouth once per day on each day of a 28-day cycle.
* Treatment will be monitored with frequent blood tests and imaging studies.
* Participants will continue to take the study drug for as long as their cancer does not worsen and side effects are not too severe.

DETAILED DESCRIPTION:
Background:

* In the United States, urothelial carcinoma (UC) of the bladder is the fourth most common malignancy in men and the ninth most common in women with an estimated 69,250 new cases and 14,990 deaths in the year 2011
* There is no Food and Drug Administration (FDA)-approved second line drug for patients with metastatic Urothelial Cancer (UC)
* Multiple lines of evidence support targeting angiogenesis in UC
* In human bladder cancer, overexpression of tyrosine-protein kinase (c-Met)/Axl/platelet derived growth factor receptor- (PDGFR)-alpha or c-Met alone showed significant correlation with poor survival
* Cabozantinib is a new chemical entity that inhibits multiple receptor tyrosine kinases with growth-promoting and angiogenic properties.
* The primary targets of cabozantinib are mesenchymal epithelial transition factor (MET), vascular endothelial factor receptor 2 (VEGFR2), and rearranged during transfection (RET)

Objectives:

- To determine the response rate of cabozantinib in patients with progressive urothelial cancer who have received prior cytotoxic chemotherapy

Eligibility:

* Patients in cohort 1 must have a histologically confirmed diagnosis of metastatic, progressive urothelial carcinoma of the bladder, urethra, ureter, or renal pelvis.
* Patients in cohort 2 must have a histologically confirmed diagnosis of bone only metastatic, urothelial carcinoma of the bladder, urethra, ureter, or renal pelvis.
* Patients in cohort 3 must have a histologically confirmed diagnosis of non-transitional cell carcinoma cancer (including but not limited to squamous cell, neuroendocrine, adenocarcinoma including urachal and sarcomatoid) of the bladder, urethra, ureter, or renal pelvis.
* Patients must have been previously treated, as defined by treatment with at least one prior cytotoxic chemotherapy regimen or agent. Patients may have received any number of prior cytotoxic agents.
* 18 years of age or older.

Design:

* A maximum of 71subjects will be enrolled in this open label, non-randomized, phase II trial of 60 mg each day of cabozantinib. Up to 50 patients will be accrued to cohort 1 (metastatic, progressive urothelial cancer. The remainder will be enrolled on exploratory cohorts 2 & 3, bone only metastatic urothelial disease and non transitional cell carcinoma (TCC) bladder cancer respectively, during the time the study is accruing patients for cohort 1. Note: Patients who tolerate cabozantinib at 60 mg daily during the first 2 cycles (first restaging time period) without (Bullet) grade 2 toxicity may undergo dose escalation to 80 mg daily at the discretion of the Principal Investigator.
* A Simon 2 stage design with alpha=0.05 and beta = 0.10 as acceptable error probabilities. Initially 21 subjects will be enrolled and followed for progression. If 2 or more of cohort 1 subjects experiences a response, enrollment will continue until a total of 41 evaluable subjects with progressive urothelial cancer have been entered. 2-3 patients per month may enroll on this trial; thus, 2 to 3 years is anticipated as the accrual period.
* Each patient will undergo response evaluation assessments with chest abdomen pelvis computed tomography (CAP CT) (or magnetic resonance imaging (MRI)) with or without 18F-Sodium Fluoride (Na18F) positron emission tomography (PET CT) every 8 weeks while on active protocol therapy starting at baseline. Patients will undergo investigational Fludeoxyglucose, (FDG) PET/CT and PET/MRI (optional) at baseline, week 4 and week 8.

ELIGIBILITY:
* INCLUSION CRITERIA:

Cohort 1 only (urothelial progressive disease)

* Patients must have a histologically confirmed diagnosis of urothelial carcinoma of the bladder, urethra, ureter, or renal pelvis. Confirmation may be obtained from any Clinical Laboratory Improvement Amendments (CLIA) certified lab.
* Patients must have progressive metastatic disease. Progressive disease will be defined as new or progressive lesions on cross-sectional imaging.
* Patients must have at least one measurable site of disease

Cohort 2 only (Bone-only)

* Patients must have a histologically confirmed diagnosis of urothelial carcinoma of the bladder, urethra, ureter, or renal pelvis. Confirmation may be obtained from any CLIA certified lab.
* Patients must not have measurable progressive disease
* Patient must have appearance of at least one new bone lesion.

Cohort 3 (Rare histologies)

* Patient must have a histologically confirmed diagnosis of non-transitional cell carcinoma of the bladder, urethra, ureter, or renal pelvis including but not limited to squamous cell, neuroendocrine, adenocarcinoma including urachal and sarcomatoid. Confirmation may be obtained from any CLIA certified lab.
* Patients must have progressive metastatic disease. Progressive disease will be defined as new or progressive lesions on cross-sectional imaging.
* Patients must have at least one measurable site of disease

All cohorts

* Patients must have been previously treated, as defined by treatment with at least one prior cytotoxic regimen or agent.
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of cabozantinib in patients <18 years of age, children are excluded from this study, but may be eligible for future pediatric trials.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2 (Karnofsky greater than or equal to 60%
* Adequate organ function as defined by the following criteria:
* Hemoglobin greater than or equal to 9 g/dL
* Absolute neutrophil count (ANC) greater than or equal to 1500/microL
* Platelets greater than or equal to 75,000/L
* Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) less than or equal to 3.0 times upper limit of normal (ULN); less than or equal to 5.0 times ULN in cases of liver metastases
* Total serum bilirubin less than or equal to 1.5 times the upper limit of normal (ULN). For subjects with known Gilberts disease or similar syndrome with slow conjugation of bilirubin, total bilirubin less than or equal to 3.0 mg/dL
* Serum creatinine less than or equal to 1.5 X institutional upper limits of normal or for patients with creatinine levels above 1.5 x institutional normal: creatinine clearance greater than or equal to 50 mL/min/1.73 m^2 by 24 hour urine collection or estimated creatinine clearance of greater than or equal to 50 mL/min. For creatinine clearance estimation , the Cockcroft and Gault equation should be used:
* Male: Creatinine Clearance (CrCl) (mL/min) = (140 - age) times wt (kg)/ (serum creatinine times 72)
* Female: Multiply above result by 0.85
* Urine protein/creatinine ratio (UPCR) less than or equal to 2
* Patient must be able to provide either archival tumor samples (haematoxylin and eosin (H&E) slides and one paraffin block or 10 unstained slides) or undergo tumor biopsy.
* Patient must be capable of understanding and complying with protocol requirements and is willing to give informed consent
* The effects of XL184 on the developing human fetus are unknown. For this reason and because tyrosine kinase inhibitors agents are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of XL184 administration.

Sexually active subjects (men and women) must agree to use medically accepted barrier methods of contraception (e.g., male or female condom) during the course of the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used. All subjects of reproductive potential must agree to use both a barrier method and a second method of birth control during the course of the study and for 4 months after the last dose of study drug(s).

- Women of childbearing potential must have a negative pregnancy test at screening. Women of childbearing potential include women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are not postmenopausal. Postmenopause is defined as amenorrhea greater than or equal to 12 consecutive months. Note: women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, ovarian suppression or any other reversible reason.

EXCLUSION CRITERIA:

* The subject has received cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) or biologic agents (eg, cytokines or antibodies) within 3 weeks, or nitrosoureas or mitomycin within 6 weeks before the first dose of study treatment.
* Prior treatment with cabozantinib
* Prior treatment with other small molecule inhibitors of Vascular Endothelial Growth Factor Receptors (VEGFR) within less than or equal to 2 years of study enrollment.
* The subject has received radiation therapy:
* to the thoracic cavity or gastrointestinal tract within 3 months before the first dose of study treatment
* to bone or brain metastasis within 14 days before the first dose of study treatment
* to any other site(s) within 28 days before the first dose of study treatment
* The subject has received radionuclide treatment within 6 weeks before the first dose of study treatment
* The subject has received prior treatment with a small molecule kinase inhibitor or a hormonal therapy (including investigational kinase inhibitors or hormones) within 14 days or five half-lives of the compound or active metabolites, whichever is longer, before the first dose of study treatment.
* The subject has received any other type of investigational agent within 28 days before the first dose of study treatment.
* The subject has not recovered to baseline or Common Terminology Criteria in Adverse Events (CTCAE). Grade 1 from toxicity due to all prior therapies except alopecia and other non-clinically significant AEs.
* The subject has a primary brain tumor
* The subject has active brain metastases, leptomeningeal or epidural disease (Note: Subjects with brain metastases previously treated with whole brain radiation or radiosurgery or subjects with epidural disease previously treated with radiation or surgery who are asymptomatic and do not require steroid treatment for at least 2 weeks before starting study treatment are eligible. Neurosurgical resection of brain metastases or brain biopsy is permitted if completed at least 3 months before starting study treatment. Baseline brain scans are not required to confirm eligibility.)
* The subject has prothrombin time (PT)/ International Normalized Ratio (INR) or partial thromboplastin time (PTT) test greater than or equal to 1.3 times the laboratory upper limit of normal (ULN) within 7 days before the first dose of study treatment.
* The subject requires treatment, in therapeutic doses, with oral anticoagulants such as warfarin prior to initiation of protocol therapy. Low dose aspirin (less than or equal to 81 mg/day), lowdose warfarin (less than or equal to 1 mg/day), and low molecular weight heparin (LMWH) are permitted. Subjects will be permitted to use anticoagulation as described if treatment is required while they are enrolled on the protocol.
* The subject requires chronic concomitant treatment of strong Cytochrome P450 3A4 (CYP3A4) inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital, and St. John's Wort).

Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/; medical reference texts such as the Physicians Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the counter medicine or herbal product.

* The subject has experienced any of the following within 3 months before the first dose of study treatment:
* clinically-significant hematemesis or gastrointestinal bleeding
* hemoptysis of greater than or equal to 0.5 teaspoon (greater than or equal to 2.5 mL) of red blood
* any other signs indicative of pulmonary hemorrhage
* The subject has tumor invading (or concern for invasion) major blood vessels
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the Investigator would make the patient inappropriate for entry into this study.
* The subject has evidence of tumor invading the gastrointestinal (GI) tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib.
* The subject is unable to swallow tablets
* The subject has a corrected Q wave, T wave (QT) interval calculated by the Fridericia formula (QTcF) >500 ms within 28 days before treatment initiation.
* The subject has a previously identified allergy or hypersensitivity to components of the study treatment formulation.
* The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.
* The subject has had within 2 years before the start of study treatment evidence of another malignancy which required systemic treatment
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with the study agents. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2012-09-11 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2020-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea B Apolo, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Thun MJ. Cancer statistics, 2009. CA Cancer J Clin. 2009 Jul-Aug;59(4):225-49. doi: 10.3322/caac.20006. Epub 2009 May 27. PMID 19474385
- [Background] McCaffrey JA, Hilton S, Mazumdar M, Sadan S, Kelly WK, Scher HI, Bajorin DF. Phase II trial of docetaxel in patients with advanced or metastatic transitional-cell carcinoma. J Clin Oncol. 1997 May;15(5):1853-7. doi: 10.1200/JCO.1997.15.5.1853. PMID 9164195
- [Background] Vaughn DJ, Broome CM, Hussain M, Gutheil JC, Markowitz AB. Phase II trial of weekly paclitaxel in patients with previously treated advanced urothelial cancer. J Clin Oncol. 2002 Feb 15;20(4):937-40. doi: 10.1200/JCO.2002.20.4.937. PMID 11844814
- [Result] Apolo AB, Nadal R, Tomita Y, Davarpanah NN, Cordes LM, Steinberg SM, Cao L, Parnes HL, Costello R, Merino MJ, Folio LR, Lindenberg L, Raffeld M, Lin J, Lee MJ, Lee S, Alarcon SV, Yuno A, Dawson NA, Allette K, Roy A, De Silva D, Lee MM, Sissung TM, Figg WD, Agarwal PK, Wright JJ, Ning YM, Gulley JL, Dahut WL, Bottaro DP, Trepel JB. Cabozantinib in patients with platinum-refractory metastatic urothelial carcinoma: an open-label, single-centre, phase 2 trial. Lancet Oncol. 2020 Aug;21(8):1099-1109. doi: 10.1016/S1470-2045(20)30202-3. Epub 2020 Jul 6. PMID 32645282
- [Derived] Folio LR, Turkbey EB, Steinberg SM, Apolo AB. Viable tumor volume: Volume of interest within segmented metastatic lesions, a pilot study of proposed computed tomography response criteria for urothelial cancer. Eur J Radiol. 2015 Sep;84(9):1708-14. doi: 10.1016/j.ejrad.2015.05.026. Epub 2015 Jun 10. PMID 26149529
- [Derived] Zuo RC, Apolo AB, DiGiovanna JJ, Parnes HL, Keen CM, Nanda S, Dahut WL, Cowen EW. Cutaneous adverse effects associated with the tyrosine-kinase inhibitor cabozantinib. JAMA Dermatol. 2015 Feb;151(2):170-7. doi: 10.1001/jamadermatol.2014.2734. PMID 25427282
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-C-0205.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 - (Urothelial Progressive Disease); Cohort 2 (Bone-only): Patients with bone-only urothelial carcinoma of the bladder, urethra, ureter, or renal pelvis.
- Cohort 3 (Rare Histologies): Patients with non-transitional cell carcinoma of the bladder, urethra, ureter, or renal pelvis.
Period: Overall Study
Arm/Group | Cohort 1 - (Urothelial Progressive Disease) | Cohort 2 (Bone-only) | Cohort 3 (Rare Histologies)
Started | 50 | 6 | 13
Completed | 42 | 5 | 10
Not Completed | 8 | 1 | 3
Not completed — Withdrawal by Subject | 5 | 1 | 1
Not completed — Adverse Event | 2 | 0 | 2
Not completed — Ineligible/Not treated | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Age, Categorical is not reported because it was not captured by cohorts.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - (Urothelial Progressive Disease) | Cohort 2 (Bone-only) | Cohort 3 (Rare Histologies) | Total
Number analyzed (Participants) | 50 | 6 | 13 | 69
Age, Continuous [Median (Full Range); unit: years] | 63 [35 to 82] | 66 [54 to 70] | 57 [22 to 74] | 63 [22 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 1 | 4 | 21
  Male | 34 | 5 | 9 | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race/Ethnicity was not captured for one participant.
  Participants
    White: number analyzed (Participants) | 49 | 6 | 13 | 68
    White | 41 | 5 | 10 | 56
    African American: number analyzed (Participants) | 49 | 6 | 13 | 68
    African American | 4 | 0 | 3 | 7
    Asian: number analyzed (Participants) | 49 | 6 | 13 | 68
    Asian | 2 | 1 | 0 | 3
    Unknown: number analyzed (Participants) | 49 | 6 | 13 | 68
    Unknown | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 50 | 6 | 13 | 69
Primary Tumor Site [Count of Participants; unit: Participants]
  Bladder | 30 | 5 | 12 | 47
  Upper tract:renal pelvis or ureter | 18 | 0 | 1 | 19
  Bladder & upper tract | 2 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Response
Description: Complete Response (CR) or Partial Response (PR) to Cabozantinib (XL184) assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.0. Complete Response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Median follow-up was 61.2 months
Population: 42/50 were analyzed in cohort 1 because 5 participants withdrew, 2 were taken off study for adverse events and 1 was ineligible. In cohort 2, 5/6 patients were analyzed because 1 withdrew; and in cohort 3, 10/13 patients were analyzed because 1 withdrew and 2 were taken off study due to adverse events.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 - (Urothelial Progressive Disease) | Cohort 2 (Bone-only) | Cohort 3 (Rare Histologies)
Number analyzed (Participants) | 42 | 5 | 10
percentage of participants | 19.1 [8.6 to 34.1] | NA [NA to NA] — The percentage and 95% CI cannot be calculated for this cohort because the participants had no measurable disease. | NA [NA to NA] — The percentage and 95% CI cannot be calculated for this cohort because the participants had no measurable disease.

2. Secondary Outcome: Overall Survival
Description: Measure the timing from the study start until death.
Time Frame: Median follow-up was 61.2 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 - (Urothelial Progressive Disease) | Cohort 2 (Bone-only) | Cohort 3 (Rare Histologies)
Number analyzed (Participants) | 42 | 5 | 10
Months | 8.1 [5.2 to 10.3] | 9.3 [4.6 to 12.5] | 5.8 [2.6 to 8.1]

3. Secondary Outcome: Progression Free Survival
Description: Measure the timing of maintaining stable disease or partial response until disease progression assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.0. Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Progressive disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions. Stable disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest um diameters while on study.
Time Frame: Median follow-up was 61.2 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 - (Urothelial Progressive Disease) | Cohort 2 (Bone-only) | Cohort 3 (Rare Histologies)
Number analyzed (Participants) | 42 | 5 | 10
Months | 3.7 [3.1 to 6.4] | 5.3 [1.8 to 8.3] | 2.9 [1.8 to 3.7]

4. Secondary Outcome: Number of Participants With Grade 4 Toxicity Hypomagnesium Related to Cabozantinib
Description: Grade 4 toxicity hypomagnesium experienced by participants related to Cabozantinib. Grade 4 toxicity is life-threatening consequences; urgent intervention indicated.
Time Frame: Median follow-up was 61.2 months
Population: We did not group the adverse events by cohort because we did not expect the cohorts to experience different adverse events as they were all getting the same medication at the same dose. And 68/69 participants were analyzed because one participant was enrolled and deemed ineligible prior to treatment.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Cohort 1 - (urothelial progressive disease) Patients with bone-only urothelial carcinoma of the bladder, urethra, ureter, or renal pelvis.
  Cohort 2 (Bone-only) Patients with bone-only urothelial carcinoma of the bladder, urethra, ureter, or renal pelvis.
  Cohort 3 (Rare histologies) Patients with non-transitional cell carcinoma of the bladder, urethra, ureter, or renal pelvis.
Arm/Group | All Participants
Number analyzed (Participants) | 68
Participants | 2

5. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Regardless of Attribution
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Median follow-up was 61.2 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 68
Participants | 67

ADVERSE EVENTS:
Time Frame: Median follow-up was 61.2 months
Description: All serious and non-serious adverse events are reported regardless of attribution. We did not group the adverse events by cohort because we did not expect the cohorts to experience different adverse events as they were all getting the same medication at the same dose. And 68/69 participants were analyzed because one participant was enrolled and deemed ineligible prior to treatment.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 66/68
Serious Adverse Events (participants affected / at risk) | 66/68
Other Adverse Events (participants affected / at risk) | 67/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=68)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3)
Alkaline phosphatase increased (Investigations) | 4 (4)
Anaphylaxis (Immune system disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Blood and lymphatic system disorders - Other, pulmonary embolus (Blood and lymphatic system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (4)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1)
Endocrine disorders - Other, thyroiditis (Endocrine disorders) | 1 (1)
Fatigue (General disorders) | 6 (6)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (6)
Hyponatremia (Metabolism and nutrition disorders) | 2 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (13)
Lipase increased (Investigations) | 1 (3)
Lymphocyte count decreased (Investigations) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — hip pain, leg pain
Nausea (Gastrointestinal disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (4)
Pain (General disorders) | 2 (5)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Platelet count decreased (Investigations) | 3 (3)
Proteinuria (Renal and urinary disorders) | 3 (3)
Rectal fistula (Gastrointestinal disorders) | 1 (1)
Serum amylase increased (Investigations) | 1 (2)
Stroke (Nervous system disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 66 (66) — Death progressive disease
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=68)
Abdominal pain (Gastrointestinal disorders) | 9 (11)
Abdominal soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 4 (6)
Alanine aminotransferase increased (Investigations) | 35 (59)
Alkaline phosphatase increased (Investigations) | 19 (28)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7)
Anal pain (Gastrointestinal disorders) | 2 (2)
Anal ulcer (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 21 (52)
Anorexia (Metabolism and nutrition disorders) | 15 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 37 (59)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (15)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (2)
Blood and lymphatic system disorders - Other, hematemesis (Blood and lymphatic system disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chills (General disorders) | 4 (4)
Concentration impairment (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 17 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Creatinine increased (Investigations) | 18 (40)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 35 (63)
Dizziness (Nervous system disorders) | 9 (11)
Dry mouth (Gastrointestinal disorders) | 5 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 9 (9)
Dysgeusia (Nervous system disorders) | 19 (20)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Edema limbs (General disorders) | 5 (5)
Endocrine disorders - Other, thyroiditis (Endocrine disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 (3)
Eye pain (Eye disorders) | 1 (2)
Fatigue (General disorders) | 28 (48)
Fever (General disorders) | 8 (9)
Flank pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Flatulence (Gastrointestinal disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Gastroparesis (Gastrointestinal disorders) | 2 (2)
Genital edema (Reproductive system and breast disorders) | 1 (1)
GGT increased (Investigations) | 4 (4)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (4)
Hematuria (Renal and urinary disorders) | 14 (14)
Hemorrhoids (Gastrointestinal disorders) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (9)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 10 (11)
Hyperthyroidism (Endocrine disorders) | 7 (8)
Hypoalbuminemia (Metabolism and nutrition disorders) | 15 (34)
Hypocalcemia (Metabolism and nutrition disorders) | 11 (36)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 4 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 13 (61)
Hyponatremia (Metabolism and nutrition disorders) | 14 (22)
Hypophosphatemia (Metabolism and nutrition disorders) | 29 (62)
Hypotension (Vascular disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 21 (27)
Infections and infestations - Other, URI (Infections and infestations) | 1 (1)
Injury, poisoning and procedural complications - Other, R. mediport (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Psychiatric disorders) | 7 (7)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Laryngitis (Infections and infestations) | 1 (1)
Lip infection (Infections and infestations) | 1 (1)
Lipase increased (Investigations) | 8 (16)
Localized edema (General disorders) | 1 (3)
Lymphocyte count decreased (Investigations) | 9 (13)
Malaise (General disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 14 (19)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — cramping - hands and legs
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 23 (26)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Neutrophil count decreased (Investigations) | 13 (23)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Oral dysesthesia (Gastrointestinal disorders) | 2 (4)
Oral pain (Gastrointestinal disorders) | 7 (7)
Pain (General disorders) | 10 (11)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 37 (77)
Palpitations (Cardiac disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 1 (1)
Paronychia (Infections and infestations) | 1 (3)
Pelvic pain (Reproductive system and breast disorders) | 3 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 33 (52)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 6 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 7 (8)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4)
Rash pustular (Skin and subcutaneous tissue disorders) | 2 (3)
Rectal fistula (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 3 (3)
Rectal pain (Gastrointestinal disorders) | 2 (2)
Rhinitis infective (Infections and infestations) | 3 (4)
Scalp pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Scrotal infection (Skin and subcutaneous tissue disorders) | 3 (4)
Scrotal pain (Reproductive system and breast disorders) | 1 (1)
Serum amylase increased (Investigations) | 8 (18)
Sinus pain (Nervous system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — hair whitening
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin infection (Infections and infestations) | 3 (3)
Skin ulceration (Skin and subcutaneous tissue disorders) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Stoma site infection (Infections and infestations) | 1 (2)
Thromboembolic event (Vascular disorders) | 4 (4)
Tooth discoloration (Gastrointestinal disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Transient ischemic attacks (Cardiac disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 4 (5)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 7 (9)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (6)
Vascular access complication (Vascular disorders) | 1 (1)
Vascular disorders - Other, L. PE (Vascular disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Vomiting (Gastrointestinal disorders) | 7 (10)
Weight loss (Investigations) | 7 (8)
White blood cell decreased (Investigations) | 22 (40)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, umbilical fungal infection (Infections and infestations) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — hands/finger cramping
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — hip pain, leg pain
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 (3) — muscle spasms
Skin and subcutaneous tissue disorders - Other, abrasion - lft. ankle (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, fever blisters on lip (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Inguinal rash (Skin and subcutaneous tissue disorders) | 1 (2)
Skin and subcutaneous tissue disorders - Other, outer stoma bleeding (Skin and subcutaneous tissue disorders) | 1 (2)
Skin and subcutaneous tissue disorders - Other, Pustule R. buttock (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Scrotal erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, Stoma ileal conduit (Skin and subcutaneous tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, thoracic muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT01688999/Prot_SAP_002.pdf
  • Informed Consent Form (2019-06-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT01688999/ICF_003.pdf